CLINICAL TRIAL: NCT02231983
Title: Clinical Characteristics and Genetic Profiles of Severe Combined Immunodeficiency in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCID-20140901
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Clinical Characteristics; Genetic Profiles
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Combined Immunodeficiency: Case histories were analyzed to grasp important characteristics of the diseases. Distribution of lymphocyte subsets from peripheral blood were examined by flow cytometry. Amplify and identify exons from gene IL-2RG by PCR and agarose gel electrophoresis, and then followed by gene sequencing.
  Interventions: Genetic: gene sequencing

INTERVENTIONS:
Genetic: gene sequencing — Amplify and identify exons from gene IL-2RG by PCR and agarose gel electrophoresis, and then followed by gene sequencing.

SUMMARY:
Severe combined immunodeficiency (SCID), a rare primary immunodeficiency dieases (PID), is poorly characterized in mainland China. We meant to explore the patients with SCID refered to our hospital and summarize their clinical manifestations and genetic features.

DETAILED DESCRIPTION:
Diagnostic criteria were based on recommendations by the Pan-American Group for Immunodeficiency and the European Society for Immunodeficiencies, which included failure to thrive, persistent diarrhea, respiratory symptoms, and oral candidiasis, or Pneumocystis pneumonia, severe bacterial infections, and disseminated Bacillus Calmette-Guérin (BCG) infection during the first 2 to 7 months of life. In addition, patients included in the study were <2 years of age, with either transplacentally acquired maternal T cells or <20 % CD3+ T cells, the absolute lymphocyte count (ALC) <3000/mm3. Exclusion criteria include HIV infection, congenital rubella, DiGeorge syndrome, Zap70 deficiency, Cartilage hair hypoplasia, PNP deficiency and MHC class II deficiency.

ELIGIBILITY:
Inclusion Criteria:

Diagnostic criteria were based on recommendations by the Pan-American Group for Immunodeficiency and the European Society for Immunodeficiencies, which included failure to thrive, persistent diarrhea, respiratory symptoms, and oral candidiasis, or Pneumocystis pneumonia, severe bacterial infections, and disseminated Bacillus Calmette-Guérin (BCG) infection during the first 2 to 7 months of life.

Exclusion Criteria: HIV infection, congenital rubella, DiGeorge syndrome, Zap70 deficiency, Cartilage hair hypoplasia, PNP deficiency and MHC class II deficiency.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: SCID patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
times of infections | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China